CLINICAL TRIAL: NCT01166282
Title: A Double-blind, Placebo-Controlled, Multicenter Study of the Efficacy and Safety of Adalimumab in Pediatric Subjects With Enthesitis Related Arthritis
Brief Title: A Study of the Efficacy and Safety of Adalimumab in Pediatric Subjects With Enthesitis Related Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M11-328; 2009-017938-46 (EudraCT Number)
Record Dates: First submitted 2010-07-19; First posted 2010-07-21 (Estimated); Results first posted 2016-06-21 (Estimated); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Enthesitis Related Arthritis (ERA)
Keywords: inflammatory back pain; ankylosing spondylitis; sacroiliitis; Juvenile Idiopathic Arthritis; enthesitis; arthritis
MeSH Terms: conditions — Arthritis, Juvenile; Spondylitis, Ankylosing; Sacroiliitis; Arthritis | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Double-blind Placebo EOW (Placebo Comparator): Placebo for adalimumab every other week (eow) for 12 weeks.
  Interventions: Biological: placebo for adalimumab
- Double-blind Adalimumab EOW (Experimental): Adalimumab (body surface area dosing 24 mg/m^2 up to a maximum of 40 mg) every other week (eow) for 12 weeks.
  Interventions: Biological: adalimumab
- Open-label Adalimumab EOW (Experimental): Adalimumab (body surface area dosing 24 mg/m^2 up to a maximum of 40 mg) every other week (eow) for up to 192 weeks.
  Interventions: Biological: adalimumab

INTERVENTIONS:
Biological: adalimumab — Adalimumab solution for subcutaneous injection.
  Other Names: ABT-D2E7; Humira
  Arms: Double-blind Adalimumab EOW; Open-label Adalimumab EOW
Biological: placebo for adalimumab — Placebo for adalimumab solution for subcutaneous injection.
  Arms: Double-blind Placebo EOW

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of adalimumab given subcutaneously every other week (eow) as compared to placebo in pediatric subjects with Enthesitis Related Arthritis (ERA).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Enthesitis Related Arthritis (ERA) as defined by International League of Associations for Rheumatology (ILAR);
* Disease activity defined as at least 3 active joints and evidence of enthesitis in at least one location;
* Inadequate response or intolerance to at least one nonsteroidal anti-inflammatory drug and at least one disease modifying anti-rheumatic drug, either sulfasalazine or methotrexate.

Exclusion Criteria:

* Any ILAR Juvenile Idiopathic Arthritis (JIA) subtype other than ERA;
* Psoriasis or a history of psoriasis in the patient or first-degree relative;
* Presence of Immunoglobulin M (IgM) rheumatoid factor;
* Presence of systemic JIA;
* History of inflammatory bowel disease;
* previous biologic therapy including anti-tumor necrosis factor (anti-TNF) therapy with a potential impact on pediatric ERA;
* Infection(s) requiring treatment with IV anti-infectives within 30 days prior to Baseline or oral anti-infectives within 14 days prior to Baseline.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2010-09; Primary Completion 2012-11 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaclyn Anderson, DO, MS, Study Director — AbbVie

REFERENCES:
- [Result] Burgos-Vargas R, Tse SM, Horneff G, Pangan AL, Kalabic J, Goss S, Unnebrink K, Anderson JK. A Randomized, Double-Blind, Placebo-Controlled Multicenter Study of Adalimumab in Pediatric Patients With Enthesitis-Related Arthritis. Arthritis Care Res (Hoboken). 2015 Nov;67(11):1503-12. doi: 10.1002/acr.22657. PMID 26223543
- [Derived] Horneff G, Seyger MMB, Arikan D, Kalabic J, Anderson JK, Lazar A, Williams DA, Wang C, Tarzynski-Potempa R, Hyams JS. Safety of Adalimumab in Pediatric Patients with Polyarticular Juvenile Idiopathic Arthritis, Enthesitis-Related Arthritis, Psoriasis, and Crohn's Disease. J Pediatr. 2018 Oct;201:166-175.e3. doi: 10.1016/j.jpeds.2018.05.042. Epub 2018 Jul 25. PMID 30054164
- See also: Related Info. — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study included a 30-day screening period.
Period: Double-blind Period
Arm/Group | Double-blind Placebo EOW | Double-blind Adalimumab EOW | Open-label Adalimumab EOW
Started | 15 | 31 | 0
Completed | 15 | 31 | 0
Not Completed | 0 | 0 | 0
Period: Open-label Period
Arm/Group | Double-blind Placebo EOW | Double-blind Adalimumab EOW | Open-label Adalimumab EOW
Started | 0 | 0 | 46
Completed | 0 | 0 | 29
Not Completed | 0 | 0 | 17
Not completed — Adverse Event | 0 | 0 | 6
Not completed — Withdrawal by Subject | 0 | 0 | 4
Not completed — Lack of Efficacy | 0 | 0 | 2
Not completed — Remission | 0 | 0 | 4
Not completed — Irregular Compliance | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population: All randomized participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Double-blind Placebo EOW | Double-blind Adalimumab EOW | Total
Number analyzed (Participants) | 15 | 31 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.9 (2.85) | 13.4 (2.86) | 12.9 (2.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 15
  Male | 9 | 22 | 31

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Number of Active Joints With Arthritis From Baseline to Week 12
Description: A joint assessment was recorded at all study visits to assess the number of active joints. A total of 72 joints were assessed for swelling not due to deformity or joints with loss of motion (LOM) plus pain and/or tenderness. Total possible scores ranges from 0 (no active joints) to 72 (all active joints). Baseline is defined as the last nonmissing value prior to the first dose of study drug. Last Observation Carried Forward (LOCF) was used for missing data.
Time Frame: Baseline and Week 12
Population: ITT population
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Double-blind Placebo EOW | Double-blind Adalimumab EOW
Number analyzed (Participants) | 15 | 31
percent change | -11.6 (100.5) | -62.6 (59.53)
Statistical Analysis 1: Comparison: Double-blind Placebo EOW vs Double-blind Adalimumab EOW; Test type: Superiority or Other; p = 0.039, ANCOVA; Mean Difference (Final Values) = -51.17, 95% CI 2-sided [-99.69 to -2.66]

2. Secondary Outcome: Number of Sites of Enthesitis: Change From Baseline to Week 12
Description: The presence of enthesitis was assessed by pressure at 35 anatomical locations. Enthesitis was classifed as either present or absent. Scores range from 0 to 35, with higher scores representing higher disease activity. Baseline is defined as the last nonmissing value prior to the first dose of study drug. LOCF was used.
Time Frame: Baseline and Week 12
Population: ITT population
Measure: Mean (Standard Deviation); unit: sites of enthesitis
Arm/Group | Double-blind Placebo EOW | Double-blind Adalimumab EOW
Number analyzed (Participants) | 15 | 31
sites of enthesitis
  Baseline | 7.8 (7.49) | 8.3 (8.89)
  Week 12 | 5.1 (8.92) | 3.9 (6.60)
  Change from Baseline to Week 12 | -2.7 (4.98) | -4.4 (6.20)
Statistical Analysis 1: Comparison: Double-blind Placebo EOW vs Double-blind Adalimumab EOW; Test type: Superiority or Other; p = 0.382, 1-way ANOVA; Mean Difference (Final Values) = -1.62, 95% CI 2-sided [-5.32 to 2.08]

3. Secondary Outcome: Tender Joint Count (TJC72): Change From Baseline to Week 12
Description: Seventy-two joints were assessed by pressure on physical examination. Joint tenderness was classified as either present or absent. Scores range from 0 to 72, with higher scores representing higher disease activity. Baseline is defined as the last nonmissing value prior to the first dose of study drug. LOCF was used.
Time Frame: Baseline and Week 12
Population: ITT population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Double-blind Placebo EOW | Double-blind Adalimumab EOW
Number analyzed (Participants) | 15 | 31
units on a scale
  Baseline | 11.9 (9.34) | 13.4 (10.49)
  Week 12 | 7.5 (8.06) | 5.5 (8.77)
  Change from Baseline to Week 12 | -4.5 (8.97) | -7.9 (8.25)
Statistical Analysis 1: Comparison: Double-blind Placebo EOW vs Double-blind Adalimumab EOW; Test type: Superiority or Other; p = 0.209, 1-way ANOVA; Mean Difference (Final Values) = -3.40, 95% CI 2-sided [-8.78 to 1.97]

4. Secondary Outcome: Swollen Joint Count (SJC68): Change From Baseline to Week 12
Description: Sixty-eight joints were assessed by physical examination. Joint swelling was classified as present or absent. Scores range from 0 to 68, with higher scores representing higher disease activity. Baseline is defined as the last nonmissing value prior to the first dose of study drug. LOCF was used.
Time Frame: Baseline and Week 12
Population: ITT population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Double-blind Placebo EOW | Double-blind Adalimumab EOW
Number analyzed (Participants) | 15 | 31
units on a scale
  Baseline | 5.2 (3.69) | 6.7 (7.30)
  Week 12 | 2.8 (2.83) | 3.2 (7.27)
  Change from Baseline to Week 12 | -2.4 (4.66) | -3.5 (5.61)
Statistical Analysis 1: Comparison: Double-blind Placebo EOW vs Double-blind Adalimumab EOW; Test type: Superiority or Other; p = 0.509, 1-way ANOVA; Mean Difference (Final Values) = -1.12, 95% CI 2-sided [-4.49 to 2.26]

5. Secondary Outcome: Percentage of Participants Achieving Pediatric American College of Rheumatology Pediatric 30% Response (ACR Pedi30)
Description: The ACR Pedi30 response is defined as ≥30% improvement in at least 3 of 6 juvenile rheumatoid arthritis (JRA) core set criteria with no more than 1 of the 6 criteria with >30% worsening. The 6 variables for the JRA core set criteria are Physician's Global Assessment (PGA) of participant's disease activity, Parent's Global Assessment of participant's overall well-being, number of active joints (joints with swelling not due to deformity or joints LOM plus pain and/or tenderness), number of joints with LOM, Childhood Health Assessment Questionnaire (CHAQ), and high sensitivity C-reactive protein (hs CRP). Baseline is the last value prior to the first dose of study drug. Non-responder imputation (NRI) was used for missing data.
Time Frame: Baseline and Week 12
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Double-blind Placebo EOW | Double-blind Adalimumab EOW
Number analyzed (Participants) | 15 | 31
percentage of participants | 60.0 | 71.0
Statistical Analysis 1: Comparison: Double-blind Placebo EOW vs Double-blind Adalimumab EOW; Test type: Superiority or Other; p = 0.514, Fisher Exact; Mean Difference (Final Values) = 11, 95% CI 2-sided [-18.5 to 40.5]

6. Secondary Outcome: Percentage of Participants Achieving Pediatric American College of Rheumatology Pediatric 50% Response (ACR Pedi50)
Description: The ACR Pedi50 response is defined as ≥50% improvement in at least 3 of 6 JRA core set criteria with no more than 1 of the 6 criteria with >30% worsening. The 6 variables for the JRA core set criteria are Physician's Global Assessment (PGA) of participant's disease activity, Parent's Global Assessment of participant's overall well-being, number of active joints (joints with swelling not due to deformity or joints LOM plus pain and/or tenderness), number of joints with LOM, Childhood Health Assessment Questionnaire (CHAQ), and high sensitivity C-reactive protein (hs CRP). Baseline is the last value prior to the first dose of study drug. NRI was used.
Time Frame: Baseline and Week 12
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Double-blind Placebo EOW | Double-blind Adalimumab EOW
Number analyzed (Participants) | 15 | 31
percentage of participants | 40.0 | 67.7
Statistical Analysis 1: Comparison: Double-blind Placebo EOW vs Double-blind Adalimumab EOW; Test type: Superiority or Other; p = 0.111, Fisher Exact; Mean Difference (Final Values) = 27.7, 95% CI 2-sided [-2.0 to 57.5]

7. Secondary Outcome: Percentage of Participants Achieving Pediatric American College of Rheumatology Pediatric 70% Response (ACR Pedi70)
Description: The ACR Pedi70 response is defined as ≥70% improvement in at least 3 of 6 JRA core set criteria with no more than 1 of the 6 criteria with >30% worsening. The 6 variables for the JRA core set criteria are Physician's Global Assessment (PGA) of participant's disease activity, Parent's Global Assessment of participant's overall well-being, number of active joints (joints with swelling not due to deformity or joints LOM plus pain and/or tenderness), number of joints with LOM, Childhood Health Assessment Questionnaire (CHAQ), and high sensitivity C-reactive protein (hs CRP). Baseline is the last value prior to the first dose of study drug. Non-responder imputation NRI was used.
Time Frame: Baseline and Week 12
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Double-blind Placebo EOW | Double-blind Adalimumab EOW
Number analyzed (Participants) | 15 | 31
percentage of participants | 20.0 | 54.8
Statistical Analysis 1: Comparison: Double-blind Placebo EOW vs Double-blind Adalimumab EOW; Test type: Superiority or Other; p = 0.031, Fisher Exact; Mean Difference (Final Values) = 34.8, 95% CI 2-sided [8.1 to 61.6]

8. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a participant which does not necessarily have a causal relationship with this treatment. A serious AE (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above. Treatment-emergent events (TEAEs or TESAE) are defined as any event that began or worsened in severity after the first dose of study drug. The investigator assessed the relationship of each event to the use of study drug as either probably related to study drug, possibly related to study drug, probably not related, or not related to study drug.
  For more details on adverse events please see the AE section below.
Time Frame: Treatment-emergent AEs (TEAEs) were collected from first dose of study drug until 70 days after the last dose of study drug (up to 212 weeks)
Population: Safety population: All randomized subjects who received at least 1 dose of study drug
Measure: Number; unit: participants
Groups:
- Any Adalimumab: All participants in this study who received at least 1 dose of adalimumab (body surface area dosing 24 mg/m^2 up to a maximum of 40 mg) every other week (double-blind or open-label) for up to 204 weeks.
Arm/Group | Double-blind Placebo EOW | Double-blind Adalimumab EOW | Any Adalimumab
Number analyzed (Participants) | 15 | 31 | 46
participants
  Any TEAE | 8 | 21 | 46
  TEAEs at least possibly related to study drug | 4 | 9 | 29
  Any severe TEAE | 0 | 0 | 7
  TESAE | 0 | 1 | 10
  Any TEAE Leading to Discontinuation of Study | 0 | 0 | 7
  Death | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent AEs (TEAEs) were collected from first dose of study drug until 70 days after the last dose of study drug (up to 212 weeks); SAEs were collected from the time informed consent was obtained (up to 216 weeks).
Description: A TEAE is defined as events with onset or worsening after the first dose of study drug to the first dose of open-label (OL) adalimumab (double blind [DB] period only), or 70 days following the last study drug administration or until the first dose of commercially available Humira after completion of the study, whichever occurs first.
Arm/Group | Double-blind Placebo EOW | Double-blind Adalimumab EOW | Any Adalimumab
Serious Adverse Events (participants affected / at risk) | 0/15 | 1/31 | 10/46
Other Adverse Events (participants affected / at risk) | 8/15 | 21/31 | 46/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind Placebo EOW (N=15) | Double-blind Adalimumab EOW (N=31) | Any Adalimumab (N=46)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 | 0 | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 1 | 1
PAIN (General disorders) | 0 | 0 | 1
APPENDICITIS (Infections and infestations) | 0 | 0 | 1
DISSEMINATED TUBERCULOSIS (Infections and infestations) | 0 | 0 | 1
PNEUMONIA (Infections and infestations) | 0 | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 0 | 0 | 1
BURNS SECOND DEGREE (Injury, poisoning and procedural complications) | 0 | 0 | 1
BURNS THIRD DEGREE (Injury, poisoning and procedural complications) | 0 | 0 | 1
CONCUSSION (Injury, poisoning and procedural complications) | 0 | 0 | 1
JOINT INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 1
TUBERCULIN TEST POSITIVE (Investigations) | 0 | 0 | 1
JOINT INSTABILITY (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
JUVENILE IDIOPATHIC ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
HEADACHE (Nervous system disorders) | 0 | 1 | 1
DIFFUSE VASCULITIS (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind Placebo EOW (N=15) | Double-blind Adalimumab EOW (N=31) | Any Adalimumab (N=46)
INCREASED TENDENCY TO BRUISE (Blood and lymphatic system disorders) | 0 | 0 | 1
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 0 | 1 | 1
EAR PAIN (Ear and labyrinth disorders) | 0 | 1 | 2
VERTIGO (Ear and labyrinth disorders) | 0 | 0 | 1
ASTIGMATISM (Eye disorders) | 0 | 0 | 1
CATARACT (Eye disorders) | 0 | 0 | 1
CONJUNCTIVITIS ALLERGIC (Eye disorders) | 0 | 0 | 2
DRY EYE (Eye disorders) | 0 | 1 | 2
VISION BLURRED (Eye disorders) | 0 | 1 | 1
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 0 | 0 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 1 | 6
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 | 2 | 2
ANAL FISSURE (Gastrointestinal disorders) | 0 | 0 | 1
CONSTIPATION (Gastrointestinal disorders) | 0 | 0 | 4
DIARRHOEA (Gastrointestinal disorders) | 0 | 1 | 8
FOOD POISONING (Gastrointestinal disorders) | 0 | 0 | 1
GASTRITIS (Gastrointestinal disorders) | 0 | 0 | 1
HAEMATOCHEZIA (Gastrointestinal disorders) | 0 | 1 | 1
NAUSEA (Gastrointestinal disorders) | 1 | 2 | 5
ODYNOPHAGIA (Gastrointestinal disorders) | 0 | 0 | 1
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 1
STOMATITIS (Gastrointestinal disorders) | 0 | 0 | 1
TOOTHACHE (Gastrointestinal disorders) | 0 | 0 | 1
VOMITING (Gastrointestinal disorders) | 0 | 1 | 4
ADVERSE DRUG REACTION (General disorders) | 0 | 1 | 2
FATIGUE (General disorders) | 0 | 0 | 1
INFLAMMATION (General disorders) | 0 | 0 | 1
INJECTION SITE ERYTHEMA (General disorders) | 0 | 1 | 3
INJECTION SITE PAIN (General disorders) | 1 | 3 | 5
INJECTION SITE PRURITUS (General disorders) | 0 | 0 | 1
INJECTION SITE URTICARIA (General disorders) | 0 | 0 | 1
NON-CARDIAC CHEST PAIN (General disorders) | 0 | 1 | 1
PAIN (General disorders) | 0 | 0 | 1
PERIPHERAL SWELLING (General disorders) | 0 | 0 | 1
PYREXIA (General disorders) | 0 | 0 | 6
HEPATOCELLULAR INJURY (Hepatobiliary disorders) | 0 | 1 | 1
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 0 | 0 | 1
ALLERGY TO ARTHROPOD BITE (Immune system disorders) | 0 | 0 | 2
ABSCESS LIMB (Infections and infestations) | 0 | 0 | 1
ACARODERMATITIS (Infections and infestations) | 1 | 0 | 0
ACUTE SINUSITIS (Infections and infestations) | 0 | 0 | 1
BRONCHITIS (Infections and infestations) | 0 | 0 | 5
BRONCHOPNEUMONIA (Infections and infestations) | 0 | 1 | 1
CANDIDA INFECTION (Infections and infestations) | 0 | 0 | 1
CELLULITIS (Infections and infestations) | 0 | 0 | 1
CONJUNCTIVITIS (Infections and infestations) | 0 | 0 | 3
CYSTITIS (Infections and infestations) | 1 | 1 | 1
EAR INFECTION (Infections and infestations) | 0 | 0 | 3
FOLLICULITIS (Infections and infestations) | 0 | 0 | 1
FUNGAL SKIN INFECTION (Infections and infestations) | 0 | 0 | 1
GASTROENTERITIS (Infections and infestations) | 0 | 2 | 8
GASTROINTESTINAL INFECTION (Infections and infestations) | 0 | 0 | 2
HERPES ZOSTER (Infections and infestations) | 0 | 0 | 2
INFLUENZA (Infections and infestations) | 0 | 0 | 2
LARYNGITIS (Infections and infestations) | 0 | 0 | 1
LATENT TUBERCULOSIS (Infections and infestations) | 0 | 0 | 1
LOCALISED INFECTION (Infections and infestations) | 0 | 0 | 1
NASOPHARYNGITIS (Infections and infestations) | 1 | 0 | 11
ORAL HERPES (Infections and infestations) | 0 | 0 | 4
ORCHITIS (Infections and infestations) | 0 | 0 | 1
OTITIS MEDIA (Infections and infestations) | 0 | 0 | 4
OTITIS MEDIA ACUTE (Infections and infestations) | 0 | 0 | 3
OTITIS MEDIA CHRONIC (Infections and infestations) | 0 | 0 | 1
PARONYCHIA (Infections and infestations) | 1 | 1 | 3
PHARYNGITIS (Infections and infestations) | 0 | 1 | 7
PHARYNGOTONSILLITIS (Infections and infestations) | 0 | 0 | 7
PILONIDAL CYST (Infections and infestations) | 0 | 0 | 1
PNEUMONIA (Infections and infestations) | 0 | 0 | 1
RASH PUSTULAR (Infections and infestations) | 0 | 0 | 1
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 3
RHINITIS (Infections and infestations) | 0 | 0 | 3
ROTAVIRUS INFECTION (Infections and infestations) | 0 | 0 | 1
SCARLET FEVER (Infections and infestations) | 0 | 0 | 1
SINUSITIS (Infections and infestations) | 0 | 1 | 5
SUBCUTANEOUS ABSCESS (Infections and infestations) | 0 | 0 | 1
TINEA INFECTION (Infections and infestations) | 0 | 0 | 1
TINEA PEDIS (Infections and infestations) | 0 | 0 | 2
TONSILLITIS (Infections and infestations) | 0 | 0 | 4
TONSILLITIS BACTERIAL (Infections and infestations) | 0 | 0 | 1
TRACHEITIS (Infections and infestations) | 0 | 0 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 3 | 16
URINARY TRACT INFECTION (Infections and infestations) | 0 | 0 | 3
VARICELLA (Infections and infestations) | 0 | 1 | 2
VIRAL INFECTION (Infections and infestations) | 0 | 0 | 3
VIRAL TONSILLITIS (Infections and infestations) | 0 | 0 | 1
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 2
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 1 | 0 | 0
CONTUSION (Injury, poisoning and procedural complications) | 0 | 0 | 2
CRANIOCEREBRAL INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 1
FALL (Injury, poisoning and procedural complications) | 0 | 0 | 2
FOOT FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 2
HAND FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 1 | 0 | 1
JOINT INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 2
LACERATION (Injury, poisoning and procedural complications) | 0 | 0 | 1
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 0 | 0 | 4
LIMB INJURY (Injury, poisoning and procedural complications) | 0 | 1 | 1
LIP INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 1
POST-TRAUMATIC PAIN (Injury, poisoning and procedural complications) | 0 | 0 | 3
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1
RIB FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 0 | 0 | 1
SKELETAL INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 1
TOOTH FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1
TRAUMATIC HAEMATOMA (Injury, poisoning and procedural complications) | 0 | 0 | 1
TRAUMATIC HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 | 1 | 1
WRIST FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 3 | 5
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 1 | 2
BLOOD PRESSURE INCREASED (Investigations) | 0 | 0 | 2
BONE DENSITY DECREASED (Investigations) | 0 | 0 | 1
HEPATIC ENZYME INCREASED (Investigations) | 0 | 1 | 3
TRANSAMINASES INCREASED (Investigations) | 0 | 0 | 1
WEIGHT INCREASED (Investigations) | 0 | 0 | 1
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1
METABOLIC SYNDROME (Metabolism and nutrition disorders) | 0 | 0 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
FOOT DEFORMITY (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
GROWING PAINS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
JUVENILE IDIOPATHIC ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 6
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
OSTEOCHONDROSIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
SYNOVIAL CYST (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
SKIN PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
DISTURBANCE IN ATTENTION (Nervous system disorders) | 0 | 0 | 1
DIZZINESS (Nervous system disorders) | 0 | 1 | 2
HEADACHE (Nervous system disorders) | 0 | 3 | 10
MIGRAINE (Nervous system disorders) | 0 | 1 | 1
PARAESTHESIA (Nervous system disorders) | 0 | 0 | 1
SYNCOPE (Nervous system disorders) | 0 | 2 | 4
TREMOR (Nervous system disorders) | 0 | 0 | 2
ANXIETY (Psychiatric disorders) | 0 | 0 | 2
ATTENTION DEFICIT/HYPERACTIVITY DISORDER (Psychiatric disorders) | 0 | 0 | 1
DEPRESSION (Psychiatric disorders) | 0 | 0 | 1
SLEEP DISORDER (Psychiatric disorders) | 0 | 1 | 2
TIC (Psychiatric disorders) | 0 | 0 | 1
BLADDER SPASM (Renal and urinary disorders) | 0 | 0 | 1
DYSURIA (Renal and urinary disorders) | 0 | 0 | 1
HAEMATURIA (Renal and urinary disorders) | 0 | 0 | 2
IGA NEPHROPATHY (Renal and urinary disorders) | 0 | 0 | 1
LEUKOCYTURIA (Renal and urinary disorders) | 0 | 0 | 1
GYNAECOMASTIA (Reproductive system and breast disorders) | 0 | 0 | 1
PENIS DISORDER (Reproductive system and breast disorders) | 0 | 0 | 1
SCROTAL PAIN (Reproductive system and breast disorders) | 0 | 0 | 1
VARICOCELE (Reproductive system and breast disorders) | 0 | 0 | 1
ADENOIDAL HYPERTROPHY (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
TONSILLAR INFLAMMATION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
VASOMOTOR RHINITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
ACNE (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
DERMATITIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
DERMATITIS ALLERGIC (Skin and subcutaneous tissue disorders) | 1 | 0 | 4
ECZEMA (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
KERATOSIS PILARIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
PITYRIASIS ROSEA (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
PSORIASIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
PUSTULAR PSORIASIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
RASH (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
SEBORRHOEIC DERMATITIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
SKIN EXFOLIATION (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
SOLAR DERMATITIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
HYPERTENSION (Vascular disorders) | 0 | 0 | 1
PREHYPERTENSION (Vascular disorders) | 0 | 0 | 1
RAYNAUD'S PHENOMENON (Vascular disorders) | 0 | 0 | 1
VASCULITIS (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.